CLINICAL TRIAL: NCT01110837
Title: Repeat Dose Nasal Allergen Challenge: Development of a Model to Investigate the Cellular and Inflammatory Changes That Occur in Allergic Rhinitis
Brief Title: Repeat Dose Nasal Allergen Challenge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: #09-3232
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis; Allergen
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Allergens

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allergen (Active Comparator)
  Interventions: Other: Allergen
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo challenge

INTERVENTIONS:
Other: Allergen — Allergen nasal challenge
  Arms: Allergen
Other: Placebo challenge — Placebo nasal challenge
  Arms: Placebo

SUMMARY:
What happens in the nose during an allergic reaction? Are there changes that a new drug could treat? What is the best way to test new drugs?The response of the nose to being exposed to cat allergen in someone who is allergic to cats. Symptoms, level of nasal blockage and cell and chemical changes that occur in the nose will be studied before and after being exposed to cat allergen. The investigators will also to see if giving repeated doses of allergen increases the response.Allergic rhinitis is a very common illness. There are over 500 million patients worldwide. It can increase the severity of associated asthma. Currently available drugs do not completely treat the symptoms. New treatments need to be found. A way of testing these drugs is very important. This study will investigate causes of the symptoms that occur in allergic rhinitis. It will also validate a proposed model to test new drugs. the Study Hypothesis is that a model of nasal allergen challenge shows an increased response (priming) with repeat challenges as determined by changes in nasal peak inspiratory flow.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged over 18 able to understand and sign the written consent form.
2. Able to comply with study procedures and protocol.
3. Positive skin prick test (wheal difference ≥ 3mm compared to negative control) to cat at or within 12 months preceding the screening visit.
4. Clear history of nasal symptoms on exposure to cats.
5. Otherwise healthy with no other health problems, other than mild asthma controlled by intermittent β2-agonist use, that may prevent the subject participating in the study.

Exclusion Criteria:

1. Presence of perennial rhinitis or seasonal allergic rhinitis.
2. TNSS < 2 at screening
3. Viral URTI within the 2 weeks prior to screening.
4. Current smoker or history of smoking within the previous 3 months.
5. Presence of any structural nasal abnormalities or nasal polyps on examination, a history of frequent nose bleeding, nasal surgery within the previous 3 months.
6. Use of concomitant medication that could affect responses to nasal challenge (e.g. corticosteroids, decongestants, anti-histamines) or any other nasally applied medication within 2 weeks prior to screening.
7. Participation in any other clinical trials within the previous 3 months.
8. Use of inhaled corticosteroids within the 2 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Change in peak nasal inspiratory flow following repeat allergen challenge | 1 year
  The peak nasal inspiratory flow will be measured using a hand-held peak flow meter, and changes will be measured following repeated allergen challenge.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Neighbour, MB BS, Principal Investigator — McMaster University
Locations (1):
- St Joseph's Healthcare, Hamitlon, Ontario, Canada